CLINICAL TRIAL: NCT03771378
Title: Efficacy and Safety of rhTPO and Eltrombopag in the Treatment of Chinese Adults With Primary Immune Thrombocytopenia (ITP):a Multicenter, Double-blind, Randomized, Controlled Trial
Brief Title: Efficacy and Safety of rhTPO and Eltrombopag in Patients With Primary Immune Thrombocytopenia (ITP)
Acronym: (ITP;rhTPO)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: The First Affiliated Hospital of Nanchang University (Other); The Third Xiangya Hospital of Central South University (Other); The First People's Hospital of Yuhang District (Other); Xiangyang Central Hospital (Other)
Responsible Party: Principal Investigator, MEI HENG, Associate Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: T18008-A
Record Dates: First submitted 2018-12-07; First posted 2018-12-11 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Primary Immune Thrombocytopenia
Keywords: ITP; rhTPO; Eltrombopag; platelets
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — eltrombopag

STUDY DESIGN:
Intervention Model Description: This study was a randomized, double-blind trial in which patients were divided into two groups, one receiving rhTPO injection and oral placebo tablet; the other group receiving oral eltrombopag and receiving a injection placebo.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Effective of rhTPO (Experimental): After enrollment, all subjects receive rhTPO, the dose is 300 U / Kg, s.c. qd, blood routine examination is detected every 3 days during treatment. If the platelet count > 250 × 109 / L, the drug will stop until the platelet count ≤ 100 × 109 / L. Efficacy and safety will be evaluated on day 15. The evaluation criteria were based on the consensus of ITP. At the same time, all subjects will receive a mimetic (tablet), po, qd.
  Interventions: Drug: rhTPO
- Effective of eltrombopag (Active Comparator): After enrollment, all subjects receive eltrombopag, the dose is 25 mg/day, po, qd, blood routine examination is detected every 3 days during treatment. If the platelet count > 250 × 109 / L, the drug will stop until the platelet count ≤ 100 × 109 / L. Efficacy and safety will be evaluated on day 15. The evaluation criteria were based on the consensus of ITP. At the same time, all subjects will give a mimetic (injection), at a dose of 300 U/Kg, s.c. qd.
  Interventions: Drug: eltrombopag

INTERVENTIONS:
Drug: rhTPO — After enrollment, all subjects receive TPO, the dose is 300 U / Kg, s.c. qd, blood routine examination is detected every 3 days during treatment. If the platelet count > 250 × 109 / L, the drug will stop until the platelet count ≤ 100 × 109 / L. Efficacy and safety will be evaluated on day 15. The evaluation criteria were based on the consensus of ITP. At the same time, all subjects will receive a mimetic (tablet), po, qd.
  Arms: Effective of rhTPO
Drug: eltrombopag — After enrollment, all subjects receive eltrombopag, the dose is 25 mg/day, po, qd. blood routine examination is detected every 3 days during treatment. If the platelet count > 250 × 109 / L, the drug will stop until the platelet count ≤ 100 × 109 / L. Efficacy and safety will be evaluated on day 15. The evaluation criteria were based on the consensus of ITP. At the same time, all subjects will give a mimetic (injection), at a dose of 300 U/Kg, s.c. qd.
  Arms: Effective of eltrombopag

SUMMARY:
Primary immune thrombocytopenia (ITP) is an acquired autoimmune hemorrhagic disease. In most cases, platelet count is negatively correlated with the severity of bleeding. Correcting low platelets is the main measure to prevent bleeding in patients with ITP. Both rhTPO and eltrombopag act on TPO receptors to increase platelets.Which one will have a better short-term (2 weeks) effect to improve platelets is the purpose of the investigator's research.

DETAILED DESCRIPTION:
Primary immune thrombocytopenia (ITP) is an acquired autoimmune hemorrhagic disease. ITP patients have an increased risk of bleeding and the clinical symptoms are petechia, ecchymosis, organ hemorrhage and even life-threatening bleeding. The mortality rate in ITP is increased approximately 60% compared with age- and sex matched comparisons, bleeding is one of the leading causes of death, thus treating and preventing bleeding is particularly important for those patients. In most cases, platelet count is negatively correlated with the severity of bleeding. Correcting low platelets is the main measure to prevent bleeding in patients with ITP. Recombinant human thrombopoietin (rhTPO), a full-length glycated TPO, is a recombinant form of c-Mpl ligand that competes with endogenous TPO for binding to TPO receptors (TPO-R, c-Mp0), many clinical trials have shown that rhTPO can efficiently and safely stimulate platelet production, increase peripheral blood platelet count. The State Food and Drug Administration approved the drug as the second-line treatment for patients with ITP in 2005. Eltrombopag is an oral, synthetic non-peptide small molecule human thrombopoietin receptor agonist approved by the US FDA in November 2008 for the treatment of patients with chronic ITP, which were inefficiently by use of glucocorticoids, immunoglobulin or splenectomy. However, pharmacokinetic study of eltrombopag showed that Asians have twice the drug exposure rate than non-Asians, so eltrombopag may have different effects in different populations. Therefore, this trial will compare the efficacy and safety of intravenous rhTPO or oral use of eltrombopag after 14 days of treatment in Chinese ITP patients.

ELIGIBILITY:
Inclusion Criteria:

1. The patient signs an informed consent form.
2. Age from 18 to 75 years old
3. The patient's first diagnosis of ITP is at least 6 months before enrollment; the platelet count must <30×109/L before taking the study drug (48 hours before).
4. Patients who were diagnosed with ITP by bone marrow biopsy and other related examinations before enrollment(Bone marrow biopsy is valid for 30 days, including 30 days);
5. The patient has been treated with splenectomy for relapse or relapse; or the patient has not undergone splenectomy, but was ineffective or relapses after treatment with at least one first line drug. Past ITP therapy can include, but is not limited to, corticosteroids, immunoglobulins (IVIG or anti-D Immunoglobulin), azathioprine, danazol, cyclophosphamide and immunomodulators;
6. Previous salvage treatments included infusion of platelets, immunoglobulins, immunomodulators, and cyclophosphamide must be completed 2 weeks prior to enrollment or treatment. Corticosteroids must end at least 14 days before enrollment.
7. Patients receiving immunosuppressive agents (including corticosteroids, azathioprine, danazol, cyclosporin A, mycophenolate mofetil) or proprietary Chinese medicines have maintained a stable therapeutic dose for at least the last month; patients who received rituximab should be discontinued half a year prior to enrollment; patients with spleen were enrolled six months after surgery;
8. No heart disease in the past 3 months, including NYHA grade III/IV charge

   , heart failure, arrhythmia or myocardial infarction requiring medical treatment;
9. Laboratory tests for coagulation function showed that prothrombin time (PT/INR) and activated partial thromboplastin time (APTT) values did not exceed 20% of the normal reference range.No history of coagulation abnormalities except ITP;
10. White blood cell count, neutrophil absolute value, hemoglobin in the normal value.Except in the following cases: a) Platelet count <30×10^9/L within Day1 or Day1 within 48 hours; b) Hemoglobin: if anemia is clearly caused by ITP (thrombocytopenia caused blood loss), the lower limit of the subject's hemoglobin level below the normal value can be based on the investigator's judgment to decide the subject whether to be selected; c) absolute neutrophil count ≥ 1.5 × 109 / L can be enrolled;
11. The following clinical biochemical indicators must be within 20% of the normal range: creatinine, alanine aminotransferase, aspartate aminotransferase, total bilirubin and alkaline phosphatase. In addition, serum albumin is not lower than the lower limit of normal value by 10%;
12. Subjects took an approved method of contraception. Female subjects (or female partners of male subjects) must be infertile (hysterectomy, bilateral salpingectomy, bilateral tubal ligation or more than 1 year after menopause) or have fertility but before the first dose for 2 weeks, study-approved contraceptive methods were used throughout the study period to 28 days after the end of the study or discontinuation of the study.Male subjects with a fertile female partner must have undergone vasectomy or consent to effective contraception throughout the study period (2 weeks prior to the first dose, throughout the study period, until the end of the study or 28 days after the discontinuation of the study) method;
13. Women with fertility must have a negative serum pregnancy test within 24 hours prior to the first dose;
14. Subjects fully understand and are able to comply with the requirements of the research protocol and are willing to complete the study as planned.

Exclusion Criteria:

1. Subjects had a history of any arterial/venous thrombosis (including stroke, transient ischemic attack, myocardial infarction, deep vein thrombosis, or pulmonary embolism) and had at least 2 of the following risk factors: hormone replacement therapy, oral contraception medicine (including estrogen), smoking, diabetes, hypercholesterolemia, drug-controlled hypertension, malignant tumors, hereditary coagulopathy;
2. Abnormalities other than ITP during the screening phase or any medical history or condition that the investigator considered unsuitable for participation in the study;
3. Patients with BMI ≥ 28;
4. Pregnant or lactating women;
5. A history of alcohol/drug abuse within 12 months prior to screening or first dose;
6. Previous treatment with a specific study drug other than rhTPO or other research treatments;
7. The subject has previously received or is currently receiving treatment with exenatide or other thrombopoietin receptor agonists;
8. Throughout the study, medications that affected platelet function (including but not limited to aspirin, clopidogrel and/or non-steroidal anti-inflammatory drugs NSAIDs) or anticoagulant therapy were continued for >3 days;
9. Accept any herbal or nutritional supplements, excluding vitamin supplements and mineral supplements within 1 week prior to the start of the study;
10. There is a history of abnormal platelet aggregation that may affect the reliability of platelet count measurements;
11. Before the first dose administration, the bone marrow biopsy showed abnormality except for ITP within 4 weeks, and the investigator judged that the abnormality made the subject unsuitable for the study, or the bone marrow biopsy showed other primary disease which caused thrombocytopenia;
12. Evidence of all laboratory or clinical HIV infections, previous clinical history of hepatitis C,hepatitis B, or active hepatitis at screening. Laboratory tests during the screening period indicate hepatitis C infection or hepatitis B infection. (Defined as HBsAg test positive, in addition, if the HBsAg test is negative, but HBcAb is positive, regardless of the status of HBsAb, HBV DNA testing is required, if positive, subjects should be excluded);
13. Rescuing treatment is required before the first dose of the drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2019-01-16 (Actual); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-05-15 (Estimated)

PRIMARY OUTCOMES:
Treatment response | 14 days from treatment
  Proportion of subjects with platelet counts ≥50×10^9/L after 14 days of treatment

SECONDARY OUTCOMES:
Remission rate | 14 days from treatment
  Complete response(platelet count ≥100 X 109/L and absence of bleeding), effective(platelet count
  ≥30X109/L and at least 2-fold increase of the baseline count and absence of bleeding), ineffective(platelet count <30 X109/L or less than 2-fold increase of the baseline platelet count or bleeding) proportion of testers after 14 days of treatment
Drug efficacy: Evaluation of effectiveness | 14 days from treatment
  During treatment, the proportion of subjects, which the platelet count at least once reached ≥50×109/L.
Evaluation of effectiveness: the proportion of subjects, which the platelet count increased at least 2 times compared with baseline | 14 days from treatment
  During treatment, the proportion of subjects, which the platelet count increased at least 2 times compared with baseline.
Using ITP-specific bleeding assessment tool (ITP-BAT) to accessvbleeding scoer | 1 month from treatment
  Bleeding manifestations were grouped into three major domains: skin (S), visible mucosae (M), and organs (O), with gradation of severity (SMOG). Each bleeding manifestation is assessed at the time of examination. Severity is graded from 0 to 3 or 4, with grade 5 for any fatal bleeding.
  Bleeding reported by the patient without medical documentation is graded 1. Within each domain, the same grade is assigned to bleeding manifestations of similar clinical impact. The "worst bleeding manifestation since the last visit" (observation period) is graded (a suitable database collection form is provided), and the highest grade within each domain is recorded.bleeding score
The incidence of adverse events | 14 days from treatment
  During treatment, the proportion of subjects, which received at least once rescue.Adverse events were evaluated according to Common Terminology Criteria for Adverse Events,version3.0,published by US National Cancer Institute.Adverse events included liver injury, fever, headache, bleeding, abdominal pain, nausea, vomiting, etc
The incidence of side effects of the drugs | 1 month from treatment
  Assessing safety through the adverse events,such as liver damage, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Hu Yu, M.D., Ph.D, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Zhou Yiming, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided
It is not clear whether the data would involve patient privacy or whether patients would agree to the disclosure of the data.

REFERENCES:
- [Result] Rodeghiero F, Stasi R, Gernsheimer T, Michel M, Provan D, Arnold DM, Bussel JB, Cines DB, Chong BH, Cooper N, Godeau B, Lechner K, Mazzucconi MG, McMillan R, Sanz MA, Imbach P, Blanchette V, Kuhne T, Ruggeri M, George JN. Standardization of terminology, definitions and outcome criteria in immune thrombocytopenic purpura of adults and children: report from an international working group. Blood. 2009 Mar 12;113(11):2386-93. doi: 10.1182/blood-2008-07-162503. Epub 2008 Nov 12. PMID 19005182
- [Result] Hodak E, David M, Ingber A, Rotem A, Hazaz B, Shamai-Lubovitz O, Sandbank M. The clinical and histopathological spectrum of IgA-pemphigus--report of two cases. Clin Exp Dermatol. 1990 Nov;15(6):433-7. doi: 10.1111/j.1365-2230.1990.tb02138.x. PMID 2279341
- [Result] Zhang Y, Kolesar JM. Eltrombopag: an oral thrombopoietin receptor agonist for the treatment of idiopathic thrombocytopenic purpura. Clin Ther. 2011 Nov;33(11):1560-76. doi: 10.1016/j.clinthera.2011.10.004. Epub 2011 Nov 4. PMID 22054810
- [Result] Erickson-Miller CL, DeLorme E, Tian SS, Hopson CB, Stark K, Giampa L, Valoret EI, Duffy KJ, Luengo JL, Rosen J, Miller SG, Dillon SB, Lamb P. Discovery and characterization of a selective, nonpeptidyl thrombopoietin receptor agonist. Exp Hematol. 2005 Jan;33(1):85-93. doi: 10.1016/j.exphem.2004.09.006. PMID 15661401
- [Result] Williams DD, Peng B, Bailey CK, Wire MB, Deng Y, Park JW, Collins DA, Kapsi SG, Jenkins JM. Effects of food and antacids on the pharmacokinetics of eltrombopag in healthy adult subjects: two single-dose, open-label, randomized-sequence, crossover studies. Clin Ther. 2009 Apr;31(4):764-76. doi: 10.1016/j.clinthera.2009.04.010. PMID 19446149
- [Result] Cheng G. Eltrombopag, a thrombopoietin- receptor agonist in the treatment of adult chronic immune thrombocytopenia: a review of the efficacy and safety profile. Ther Adv Hematol. 2012 Jun;3(3):155-64. doi: 10.1177/2040620712442525. PMID 23556122
- [Result] Tomiyama Y, Miyakawa Y, Okamoto S, Katsutani S, Kimura A, Okoshi Y, Ninomiya H, Kosugi H, Nomura S, Ozaki K, Ikeda Y, Hattori T, Katsura K, Kanakura Y. A lower starting dose of eltrombopag is efficacious in Japanese patients with previously treated chronic immune thrombocytopenia. J Thromb Haemost. 2012 May;10(5):799-806. doi: 10.1111/j.1538-7836.2012.04695.x. PMID 22409309
- [Derived] Mei H, Xu M, Yuan G, Zhu F, Guo J, Huang R, Qin J, Lv T, Qin F, Cai H, Yin P, Qin T, Hu Y. A multicentre double-blind, double-dummy, randomised study of recombinant human thrombopoietin versus eltrombopag in the treatment of immune thrombocytopenia in Chinese adult patients. Br J Haematol. 2021 Dec;195(5):781-789. doi: 10.1111/bjh.17808. Epub 2021 Sep 16. PMID 34528239

DOCUMENTS (1):
  • Informed Consent Form (2018-12-16): https://cdn.clinicaltrials.gov/large-docs/78/NCT03771378/ICF_000.pdf